CLINICAL TRIAL: NCT05710796
Title: AN OBSERVATIONAL STUDY ON CARDIOVASCULAR INVOLVEMENT IN COVID RECOVERED PATIENTS
Status: Completed | Type: Observational
Sponsor: Kakatiya University (Other)
Responsible Party: Principal Investigator, Satyam Suman, Department of Pharmacy Practice, Kakatiya University
Other Study IDs: IECHS/CCP/DOPP/09/04
Record Dates: First submitted 2023-01-30; First posted 2023-02-02 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-02

CONDITIONS: Gender Discrimination; Cardiac Event; Complication
Keywords: Cardiovascular involvement; COVID 19 disease; Gender difference
MeSH Terms: conditions — Sexism; Cardiovascular Diseases | interventions — Sex

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- All population: The total population reported to Cardiology department during enrollment period
  Interventions: Behavioral: Difference in gender, response to disease, diagnostic test values
- COVID recovered: Patient having history of COVID 19 disease
  Interventions: Behavioral: Difference in gender, response to disease, diagnostic test values
- No history of COVID: Population those who never exposed to COVID 19 disease and never suffers
  Interventions: Behavioral: Difference in gender, response to disease, diagnostic test values

INTERVENTIONS:
Behavioral: Difference in gender, response to disease, diagnostic test values — Gender difference: Prevalence of disease in male vs female Response to disease: Which group is more prone to cardiac involvement Diagnostic tests: Diagnostic confirmation of disease

SUMMARY:
Aim of the study is to evaluate the prevalence and bring awareness ofcardiovascular complications in COVID-19 recovered patients. Study is conducted at single site, which is Srinivasa Heart Centre, Warangal, Telangana state in India for the duration of 4 months. The sample size is calculated 500 patients and the study is cohort, observational study. Patient consent has been taken before enrolment.

DETAILED DESCRIPTION:
The aim of the study is to evaluate the prevalence and bring awareness of cardiovascular complications in COVID-19 recovered patients.

Objectives of the study:

1. To study causes and risk factors of cardiac disorders associated with COVID-19
2. To identify different types of cardiac symptoms patients, present with
3. To study the impact of co-morbidities on COVID-19 recovered patients
4. To study treatment patterns and duration of therapy

Plan to study:

* To select the patient based on inclusion and exclusion criteria
* To collect the patient information from case sheets and by patient interaction
* To identify different types of cardiac disorders related to COVID-19 or its treatment regimen
* To study the management of COVID-19 complication and related cardiovascular disorders

Study Sites: Srinivasa Heart Centre, Warangal (T.S) Study Design: Observational cohort study Study Duration: 4 months

Subject Eligibility:

1. Inclusion Criteria

   * Patients who are willing to participate
   * Patients having previous COVID-19 treatment record
   * Prescriptions reported during the study period
   * The prescription which is legible and complete
2. Exclusion Criteria

   * Patients who are not willing to participate
   * The patient having no history of COVID-19 and available data

Source of the data:

1. Review of patient case sheet, prescription and lab reports
2. Personal interaction with patients and caregivers

Sample size: 500 Patients

ELIGIBILITY:
Inclusion Criteria:

* Patients who are willing to participate
* Patients having previous COVID-19 treatment record
* Prescriptions reported during the study period
* The prescription which is legible and complete

Exclusion Criteria:

* Patients who are not willing to participate
* The patient having no history of COVID-19 and available data

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient reporting to the cardiology department during study period
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-04-29 (Actual)

PRIMARY OUTCOMES:
ECG, Lipid profile, TMT, and 2D Echo | September 2021 to February 2022
  The following tests are performed to every individuals and relevant report are considered

CONTACTS AND LOCATIONS:
Locations (1):
- Srinivasa Heart Centre, Warangal, Telangana, India

IPD SHARING:
Plan to Share IPD: Undecided
May be in future it will be needed